CLINICAL TRIAL: NCT00711178
Title: A Randomized Multicenter Study of Daylight Mediated Photodynamic Therapy (PDT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Professor Hans Christian Wulf, Department of Dermatology, Bispebjerg Hospital, Denmark, Bispebjerg Hospital, University of Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Multicenter Sun-PDT
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2008-03

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 2 hours sunlight
  Interventions: Procedure: Photodynamic therapy with methyl aminolevulinate
- B (Active Comparator): 3 hours of sunlight
  Interventions: Procedure: Photodynamic therapy with methyl aminolevulinate

INTERVENTIONS:
Procedure: Photodynamic therapy with methyl aminolevulinate — daylight mediated photodynamic therapy

SUMMARY:
A randomised, multi-center study of daylight mediated photodynamic therapy (PDT) with Metvix in patients with multiple actinic keratosis on the face and/or scalp.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, 5 AK in face and scalp

Exclusion Criteria:

* immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
response rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark